CLINICAL TRIAL: NCT02188303
Title: A Single and Multiple Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of the Oxyntomodulin Analog, LY2944876, in Healthy Japanese Subjects and Healthy Non-Japanese Subjects
Brief Title: A Study of LY2944876 in Healthy Japanese and Non-Japanese Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The termination criteria of the protocol was met during dose escalation.
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 15247; I7I-EW-XNAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Single Dose, Cohorts 1-3) (Placebo Comparator): Single dose of placebo matching LY2944876 administered subcutaneous (SC) on Day 1
  Interventions: Drug: Placebo
- LY2944876 (Single Dose, Cohorts 1-3) (Experimental): Single dose of 10 milligrams (mg) of LY2944876 administered SC on Day 1
  Interventions: Drug: LY2944876
- Placebo (Multiple Dose, Cohort 4) (Placebo Comparator): Placebo matching LY2944876 administered once daily SC on Days 1-7
  Interventions: Drug: Placebo
- LY2944876 (Multiple Dose, Cohort 4) (Experimental): 40 mg LY2944876 administered once daily SC on Days 1-7
  Interventions: Drug: LY2944876
- Placebo (Multiple, Cohort 5) (Placebo Comparator): Placebo matching LY2944876 administered once daily SC on Days 1, 4, 6, 8, 10 and 12
  Interventions: Drug: Placebo
- LY2944876 (Multiple Dose, Cohort 5, Titrated) (Experimental): LY2944876 in titrated doses of 15 mg on Day 1, 30 mg on Day 4, up to 60 mg on Day 6, and up to 80 mg on Days 8, 10 and 12 administered once daily SC
  Interventions: Drug: LY2944876

INTERVENTIONS:
Drug: LY2944876 — Administered SC
  Arms: LY2944876 (Multiple Dose, Cohort 4); LY2944876 (Multiple Dose, Cohort 5, Titrated); LY2944876 (Single Dose, Cohorts 1-3)
Drug: Placebo — Administered SC
  Arms: Placebo (Multiple Dose, Cohort 4); Placebo (Multiple, Cohort 5); Placebo (Single Dose, Cohorts 1-3)

SUMMARY:
LY2944876 is an investigative drug for the treatment of Type 2 Diabetes Mellitus. Part A of the study will assess the safety and tolerability of single doses of LY2944876 in Japanese participants. Participation is expected to last up to about 7 weeks, not including screening.

Part B of the study will investigate the safety and tolerability of multiple doses of LY2944876 in non Japanese participants. Participation is expected to last up to about 8 weeks, not including screening.

All doses will be administered as injections into the fatty layer just beneath the skin.

Screening is required within 28 days prior to the start of the study. All participants will attend a post study safety assessment approximately 6 weeks after their final dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or female participants
* Are first generation Japanese participants (Part A) or non-Japanese participants (Part B)
* Have a body mass index (BMI) of 18.5 to 30 kilogram per meter square (kg/m^2), inclusive, for Part A and a BMI of 25 to 40 kg/m^2, inclusive, for Part B at screening
* Have normal blood pressure and heart rate (after approximately 5 minutes supine and approximately 2 minutes standing) as determined by the investigator at screening

Exclusion Criteria:

* Have known allergies to LY2944876, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening and/or baseline that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history of acute or chronic pancreatitis or elevation in serum lipase and/or amylase greater than 2 times the upper limit of normal (ULN) at screening and/or baseline
* Have known or ongoing psychiatric disorders considered clinically significant in the opinion of the investigator
* Have undergone any form of bariatric surgery
* Have fasting blood glucose levels greater than or equal to (≥) 7 millimoles per liter (mmol/L) [≥126 milligrams per deciliter (mg/dL)] at screening
* Have fasting triglycerides levels ≥300 mg/dL (3.4 mmol/L) at screening
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or an alanine transaminase (ALT) or aspartate aminotransferase (AST) levels greater than (>) 2.5 times the ULN at screening and/or baseline
* Have used or intend to use medications that promote weight loss, within 3 months prior to screening, for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A / Cohorts 1-3 - Placebo: Placebo, Single Dose Administered Subcutaneously (SC) on Day 1
- Part A / Cohort 1 - 10 mg LY2944876: 10 milligram (mg) LY2944876, Single Dose Administered SC on Day 1
- Part A / Cohort 2 - 30 mg LY2944876: 30 mg LY2944876, Single Dose Administered SC on Day 1
- Part A / Cohort 3 - 50 mg LY2944876: 50 mg LY2944876, Single Dose Administered SC on Day 1
- Part B / Cohort 4 - Placebo: Placebo Administered Once Daily (QD) SC, Days 1-7
- Part B / Cohort 4 - 40 mg LY2944876: 40 mg LY2944876 Administered QD SC, Days 1-7
- Part B / Cohort 5 - Placebo: Placebo Administered QD SC, Day 1, 4 and 6.
- Part B / Cohort 5 - 15-60 mg Titrated LY2944876: LY2944876 Administered QD SC 15 mg on Day 1, 30 mg on Day 4 and up to 60 mg on Day 6.
Period: Overall Study
Arm/Group | Part A / Cohorts 1-3 - Placebo | Part A / Cohort 1 - 10 mg LY2944876 | Part A / Cohort 2 - 30 mg LY2944876 | Part A / Cohort 3 - 50 mg LY2944876 | Part B / Cohort 4 - Placebo | Part B / Cohort 4 - 40 mg LY2944876 | Part B / Cohort 5 - Placebo | Part B / Cohort 5 - 15-60 mg Titrated LY2944876
Started | 6 | 6 | 6 | 6 | 4 | 12 | 2 | 6
Completed | 6 | 6 | 6 | 6 | 4 | 10 | 0 (Protocol-defined dose termination criteria met, dosing stopped on Day 5 and study was terminated.) | 0 (Protocol-defined dose termination criteria met, dosing stopped on Day 5 and study was terminated.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Not completed — Dose Termination Criteria Met | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Part A / Cohorts 1-3 - Placebo: Placebo, Single Dose Administered SC
- Part A / Cohort 1 - 10 mg LY2944876: LY2944876 10 mg, Single Dose Administered SC
- Part A / Cohort 2 - 30 mg LY2944876: LY2944876 30 mg, Single Dose Administered SC
- Part A / Cohort 3 - 50 mg LY2944876: LY2944876 50 mg, Single Dose Administered SC
- Part B / Cohort 4 - Placebo: Placebo Administered QD SC, Days 1-7
- Part B / Cohort 4 - 40 mg LY2944876: LY2944876 40 mg, Administered QD SC, Days 1-7
- Part B / Cohort 5 - Placebo: Placebo, Administered QD SC, Days 1, 4 and 6.
- Total: Total of all reporting groups
Arm/Group | Part A / Cohorts 1-3 - Placebo | Part A / Cohort 1 - 10 mg LY2944876 | Part A / Cohort 2 - 30 mg LY2944876 | Part A / Cohort 3 - 50 mg LY2944876 | Part B / Cohort 4 - Placebo | Part B / Cohort 4 - 40 mg LY2944876 | Part B / Cohort 5 - Placebo | Part B / Cohort 5 - 15-60 mg Titrated LY2944876 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 12 | 2 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age data was presented per Cohort (Part A and Part B).
  Years
    Cohorts 1-3: number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 24
    Cohorts 1-3 | 29.2 (5.4) | 33.2 (5.8) | 29.5 (3.9) | 29.2 (3.5) |  |  |  |  | 30.3 (4.8)
    Cohorts 4-5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 12 | 2 | 6 | 24
    Cohorts 4-5 |  |  |  |  | 47.5 (18.2) | 46.3 (16.4) | 56.5 (7.8) | 46.3 (16.6) | 47.3 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 8
  Male | 6 | 6 | 6 | 6 | 2 | 9 | 1 | 4 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 6 | 6 | 6 | 0 | 1 | 0 | 0 | 25
  White | 0 | 0 | 0 | 0 | 4 | 11 | 2 | 6 | 23
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 6 | 6 | 6 | 6 | 4 | 12 | 2 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to Be Related to Study Drug Administration
Description: An SAE is any adverse event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. The number of participants with 1 or more SAEs considered by the investigator to be related to study drug administration is reported. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, were reported in the Reported Adverse Events module.
Time Frame: Pre-dose (PRD) through Study Completion (Up to Day 40)
Population: All enrolled participants, whether or not they completed all protocol requirements.
Measure: Number; unit: Participants
Groups:
- Cohorts 1-3 - Placebo: Placebo, Single Dose Administered SC
- Cohort 1 - 10 mg LY2944876: 10 mg LY2944876, Single Dose Administered SC
- Cohort 2 - 30 mg LY2944876: 30 mg LY2944876, Single Dose Administered SC
- Cohort 3 - 50 mg LY2944876: 50 mg LY2944876, Single Dose Administered SC
- Cohort 4 - Placebo: Placebo Administered QD SC, Days 1-7
- Cohort 4 - 40 mg LY2944876: 40 mg LY2944876 Administered QD SC, Days 1-7
- Cohort 5 - Placebo: Placebo Administered QD SC, Day 1, Day 4 and Day 6.
- Cohort 5 - 15-60 mg Titrated LY2944876: LY2944876 Administered QD SC 15 mg on Day 1, 30 mg on Day 4 and up to 60 mg on Day 6.
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - 10 mg LY2944876 | Cohort 2 - 30 mg LY2944876 | Cohort 3 - 50 mg LY2944876 | Cohort 4 - Placebo | Cohort 4 - 40 mg LY2944876 | Cohort 5 - Placebo | Cohort 5 - 15-60 mg Titrated LY2944876
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 12 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve - Time Zero to 168 Hours Post-dose [AUC(0-168h)] of LY2944876
Time Frame: Cohorts1-3:Day1 PRD,8,12,24,32,48,56,72,96,168Hrs;Days15,28,42:Cohort4:Day1 PRD,12 Hrs;Days2,3,4,5,6 PRD;Day7 PRD,12,24,36,48,56,72,96,168 Hrs;Days21,34,49: Cohort 5:Day1 PRD,12,24,48 Hrs;Days4,6,8,10 PRD;Day12 PRD,12,24,36,48,56,72,96,168 Hrs;Day26,39,53
Population: All randomized participants receiving at least one dose of the investigational product and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms∙hours/milliliters (ng∙h/mL)
Groups:
- Cohort 4 - 40 mg LY2944876: 40 mg LY2944876 Administered QD SC, Day 7
- Cohort 5 - 15-60 mg Titrated LY2944876: LY2944876 Administered QD SC, titrated up to 60 mg on Day 6
Arm/Group | Cohort 1 - 10 mg LY2944876 | Cohort 2 - 30 mg LY2944876 | Cohort 3 - 50 mg LY2944876 | Cohort 4 - 40 mg LY2944876 | Cohort 5 - 15-60 mg Titrated LY2944876
Number analyzed (Participants) | 6 | 6 | 6 | 10 | 5
nanograms∙hours/milliliters (ng∙h/mL) | 105000 (32) | 307000 (38) | 495000 (34) | 1789000 (15) | 803000 (24)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2944876
Time Frame: as for outcome 2
Population: All randomized participants receiving at least one dose of the investigational product and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Cohort 3 - LY2944876 50 mg: 50 mg LY2944876, Single Dose Administered SC
Arm/Group | Cohort 1 - 10 mg LY2944876 | Cohort 2 - 30 mg LY2944876 | Cohort 3 - LY2944876 50 mg | Cohort 4 - 40 mg LY2944876 | Cohort 5 - 15-60 mg Titrated LY2944876
Number analyzed (Participants) | 6 | 6 | 6 | 10 | 5
nanograms/milliliter (ng/mL) | 790 (33) | 2360 (36) | 3640 (35) | 11700 (26) | 5470 (22)

ADVERSE EVENTS:
Groups:
- Cohorts 1-3 - Placebo: Placebo, Single Dose Administered Subcutaneously (SC)
- Cohort 1 - LY2944876 10 mg: LY2944876 10 mg, Single Dose Administered SC
- Cohort 2 - LY2944876 30 mg: LY2944876 30 mg, Single Dose Administered SC
- Cohort 3 - LY2944876 50 mg: LY2944876 50 mg, Single Dose Administered SC
- Cohort 4 - LY2944876 40 mg: LY2944876 40 mg Administered QD SC, Days 1-7
- Cohort 5 - Placebo: Placebo Administered QD SC, Day 1, Day 4, and Day 6.
- Cohort 5 - 15-80 mg Titrated LY2944876: LY2944876 Administered QD SC 15 mg on Day 1, 30 mg on Day 4 and up to 60 mg on Day 6.
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - LY2944876 10 mg | Cohort 2 - LY2944876 30 mg | Cohort 3 - LY2944876 50 mg | Cohort 4 - Placebo | Cohort 4 - LY2944876 40 mg | Cohort 5 - Placebo | Cohort 5 - 15-80 mg Titrated LY2944876
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/12 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 4/6 | 6/6 | 4/4 | 12/12 | 2/2 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1-3 - Placebo (N=6) | Cohort 1 - LY2944876 10 mg (N=6) | Cohort 2 - LY2944876 30 mg (N=6) | Cohort 3 - LY2944876 50 mg (N=6) | Cohort 4 - Placebo (N=4) | Cohort 4 - LY2944876 40 mg (N=12) | Cohort 5 - Placebo (N=2) | Cohort 5 - 15-80 mg Titrated LY2944876 (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 6 (6) | 1 (1) | 5 (5)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 8 (8) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 9 (9) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days